CLINICAL TRIAL: NCT01536145
Title: An Open Label Phase I Study Of CP-751,871 In Patients With Multiple Myeloma
Brief Title: CP-751,871 Treatment For Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4021001
Record Dates: First submitted 2012-02-14; First posted 2012-02-20 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Multiple Myeloma
Keywords: IGF-1R inhibitor; CP-751871; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — figitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single agent CP-751,871 (Experimental): dose escalation design
  Interventions: Drug: CP-751,871

INTERVENTIONS:
Drug: CP-751,871 — CP-751,871 was given at doses ranging from 0.025 mg/kg up to 20 mg/kg IV every 4 weeks until disease progression or lack of tolerability

SUMMARY:
This study represents the first-in-human study for CP-751,871. The study aimed to define the safety, tolerability, and maximum tolerated dose of CP-751,871 in patients with multiple myeloma through a dose escalation design.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated multiple myeloma with a quantifiable serum (M spike ≥ 1 g/dL) and/or urine (≥ 200 mg/24-hr) paraprotein
* Adequate bone marrow, renal, liver and cardiac function
* Eastern Cooperative Oncology Group [ECOG] performance status less than or equal to 2

Exclusion Criteria:

* Prior allogeneic stem cell transplant (alloSCT)
* Myelosuppressive chemotherapy or immunotherapy within 3 weeks prior to treatment with CP-751,871
* Prior organ allograft
* Concurrent use of insulin, oral hypoglycemic medication, growth hormone (GH), or growth hormone inhibitors
* Female patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2003-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, New York, New York

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021001&StudyName=CP-751%2C871%20Treatment%20For%20Patients%20With%20Multiple%20Myeloma%20

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-751,871 0.025 mg/kg: CP-751,871 0.025 milligram/kilogram (mg/kg) administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks)
- CP-751,871 0.05 mg/kg: CP-751,871 0.05 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks)
- CP-751,871 0.1 mg/kg: CP-751,871 0.1 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks)
- CP-751,871 0.2 mg/kg: CP-751,871 0.2 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks)
- CP-751,871 0.4 mg/kg: CP-751,871 0.4 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks)
- CP-751,871 0.8 mg/kg: CP-751,871 0.8 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks)
- CP-751,871 1.5 mg/kg: CP-751,871 1.5 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks)
- CP-751,871 3 mg/kg: CP-751,871 3 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent Cycles, starting from Cycle 2 (4 weeks)
- CP-751,871 6 mg/kg: CP-751,871 6 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks)
- CP-751,871 10 mg/kg: CP-751,871 10 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks) and subsequent cycles, starting from Cycle 2 (4 weeks)
- CP-751,871 20 mg/kg: CP-751,871 20 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks) and subsequent cycles, starting from Cycle 2 (4 weeks)
Period: Overall Study
Arm/Group | CP-751,871 0.025 mg/kg | CP-751,871 0.05 mg/kg | CP-751,871 0.1 mg/kg | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Started | 3 | 4 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 7 | 10
Completed | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Not Completed | 3 | 4 | 2 | 2 | 2 | 3 | 2 | 4 | 3 | 6 | 10
Not completed — Progressive disease | 3 | 4 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- CP-751,871: CP-751,871 0.025, 0.05, 0.1, 0.2, 0.4, 0.8, 1.5, 3 and 6 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks); CP-751,871 10 and 20 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks) and subsequent cycles, starting from Cycle 2 (4 weeks)
Arm/Group | CP-751,871
Number analyzed (Participants) | 47
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The highest dose level at which not more than 1 dose-limiting toxicity (DLT) was observed during Cycle 1 in 6 participants
Time Frame: Baseline up to Cycle 1 (Week 4 or Week 8)
Population: All participants who received at least 1 dose of study drug CP-751,871.
Measure: Number; unit: mg/kg
Groups:
- CP-751,871 0.025-20 mg/kg: CP-751,871 0.025, 0.05, 0.1, 0.2, 0.4, 0.8, 1.5, 3 and 6 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks); CP-751,871 10 and 20 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks) and subsequent cycles, starting from Cycle 2 (4 weeks)
Arm/Group | CP-751,871 0.025-20 mg/kg
Number analyzed (Participants) | 47
mg/kg | NA — CP-751,871 was safe and well tolerated at dose levels up to 20 mg/kg, and MTD was not achieved.

2. Secondary Outcome: Single Dose End-of-infusion Concentration (Cinf) for CP-751,871
Time Frame: 1 hour postdose in Cycle 1
Population: All participants treated who had at least 1 concentration.
Measure: Mean (Standard Deviation); unit: milligram/liter (mg/L)
Arm/Group | CP-751,871 0.025 mg/kg | CP-751,871 0.05 mg/kg | CP-751,871 0.1 mg/kg | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 4 | 2 | 3 | 4 | 3 | 7 | 9
milligram/liter (mg/L) | 0 (NA) — Number of participants analyzed was less than 3, thus standard deviation was not calculated. | 0.381 (0.448) | 5.32 (6.85) | 5.36 (1.52) | 6.66 (2.84) | 14.6 (NA) — Number of participants analyzed was less than 3, thus standard deviation was not calculated. | 26.0 (9.03) | 62.7 (13.5) | 159 (57.2) | 165 (57.3) | 238 (215)

3. Secondary Outcome: Single Dose Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for CP-751,871
Time Frame: Cycle 1: predose; 1; 24; 48; 72; 168; 336; 504, 672 and 1008 (for participants with an up to 8-week Cycle 1 only) hours postdose
Population: All participants treated who had at least 1 of the pharmacokinetic (PK) parameters of primary interest.
Measure: Mean (Standard Deviation); unit: milligram•hour/liter (mg•hr/L)
Arm/Group | CP-751,871 0.1 mg/kg | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 2 | 3 | 4 | 3 | 3 | 4 | 3 | 7 | 6
milligram•hour/liter (mg•hr/L) | 101 (NA) — Number of participants analyzed was less than 3, thus standard deviation was not calculated. | 202 (29.2) | 1016 (583) | 2079 (1413) | 8380 (4533) | 15436 (6406) | 26144 (2672) | 38700 (15019) | 95565 (25891)

4. Secondary Outcome: Single Dose Volume of Distribution (Vz) for CP-751,871
Time Frame: Cycle 1: predose; 1; 24; 48; 72; 168; 336; 504 and 672 and 1008 (for participants with an up to 8-week Cycle 1 only) hours postdose
Population: All participants treated who had at least 1 of the PK parameters of primary interest.
Measure: Mean (Standard Deviation); unit: milliliter/kilogram (mL/kg )
Arm/Group | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 2 | 3 | 3 | 5
milliliter/kilogram (mL/kg ) | 46.3 (12.2) | 63.3 (26.4) | 64.5 (29.7) | 52.0 (NA) — Number of participants analyzed was less than 3, thus standard deviation was not calculated. | 90.0 (18.2) | 81.9 (28.5) | 93.0 (14.3)

5. Secondary Outcome: Single Dose Plasma Decay Half-life (t1/2) for CP-751,871
Time Frame: as for outcome 4
Population: All participants treated who had at least 1 of the PK parameters of primary interest.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 2 | 3 | 3 | 5
days | 1.70 (0.631) | 4.63 (2.88) | 4.10 (0.0566) | 9.15 (NA) — Number of participants analyzed was less than 3, thus standard deviation was not calculated. | 12.7 (1.59) | 12.7 (4.61) | 12.1 (3.42)

6. Secondary Outcome: Single Dose Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] for CP-751,871
Time Frame: as for outcome 4
Population: All participants treated who had at least 1 of the PK parameters of primary interest.
Measure: Mean (Standard Deviation); unit: mg•hr/L
Arm/Group | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 2 | 3 | 3 | 5
mg•hr/L | 249 (42.5) | 1121 (645) | 2191 (1396) | 11035 (NA) — Number of participants analyzed was less than 3, thus standard deviation was not calculated. | 15025 (3673) | 32360 (4023) | 46275 (16606)

7. Secondary Outcome: Single Dose Volume of Distribution at Steady State (Vss) for CP-751,871
Time Frame: as for outcome 4
Population: All participants treated who had at least 1 of the PK parameters of primary interest.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 2 | 3 | 3 | 5
mL/kg | 46.0 (11.9) | 65.9 (24.7) | 72.6 (21.1) | 50.9 (NA) — Number of participants analyzed was less than 3, thus standard deviation was not calculated. | 81.4 (16.6) | 69.4 (16.0) | 92.1 (15.8)

8. Secondary Outcome: Single Dose Systemic Clearance (CL) for CP-751,871
Time Frame: as for outcome 4
Population: All participants treated who had at least 1 of the PK parameters of primary interest.
Measure: Mean (Standard Deviation); unit: milliliter/day/kilogram (mL/day/kg)
Arm/Group | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 2 | 3 | 3 | 5
milliliter/day/kilogram (mL/day/kg) | 19.7 (3.65) | 11.9 (8.75) | 10.9 (5.09) | 3.57 (NA) — Number of participants analyzed was less than 3, thus standard deviation was not calculated. | 4.98 (1.14) | 4.50 (0.602) | 5.71 (1.83)

9. Secondary Outcome: Multiple Dose Cinf for CP-751,871
Time Frame: 1 hour postdose in Cycles 2 up to 16
Population: Multiple dose Cinf data were listed for individual subjects, however were not summarized by descriptive statistics.
Arm/Group | CP-751,871 0.025 mg/kg | CP-751,871 0.05 mg/kg | CP-751,871 0.1 mg/kg | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Multiple Dose Minimum Observed Plasma Trough Concentration (Cmin) for CP-751,871
Time Frame: 0 hour (predose) in Cycles 2 up to 16
Population: Multiple dose Cmin data were listed for individual subjects, however were not summarized by descriptive statistics.
Arm/Group | CP-751,871 0.025 mg/kg | CP-751,871 0.05 mg/kg | CP-751,871 0.1 mg/kg | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Pharmacodynamic-based Dose
Description: The dose associated with PK exposure that was associated with 80% of the maximal effect based on down-regulation of insulin-like growth factor 1 receptor (IGF-1R) expression
Time Frame: Cycle 1 (Week 4 or Week 8)
Population: Data from analysis of the PK/pharmacodynamic relationship could not permit a reliable estimate of the pharmacodynamic-based dose.
Arm/Group | CP-751,871 0.025-20 mg/kg
Number analyzed (Participants) | 0

12. Secondary Outcome: Human Anti-human Antibody (HAHA) Response to CP-751,871
Time Frame: 30 minutes predose in Cycle 1 and subsequent cycles, end of study visit (Days 30 and 60) for dose levels below 0.8 mg/kg; 30 minutes predose in Cycle 1 and last scheduled follow-up visit for dose levels greater than or equal to 0.8 mg/kg
Population: All treated participants with HAHA samples collected at time points when circulating CP-751,871 concentrations were below the lower limit of quantification.
Measure: Number
Arm/Group | CP-751,871 0.025-20 mg/kg
Number analyzed (Participants) | 28
Value | NA — None of the analyzed samples were positive for anti-CP-751,871 antibodies, as suggested by a titer measurement of less than 3.32.

13. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based on assessment of confirmed complete remission (CR) or confirmed partial remission (PR) according to Southwest Oncology Group (SWOG) criteria. CR were those with absence of bone marrow or blood findings of multiple myeloma. PR were those with a 50-74% reduction in the quantitative immunoglobulin, and if present, a 50-89% reduction in the urine M-component (Bence-Jones protein).
Time Frame: Baseline, Day 1 at predose/cycle, end of study (30-60 days post last dose)
Population: All participants who completed a minimum of 1 cycle of treatment were evaluable for response. Participants who developed early progressive disease (regardless of the duration of study treatment) prior to response evaluation were also evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | CP-751,871 0.025 mg/kg | CP-751,871 0.05 mg/kg | CP-751,871 0.1 mg/kg | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 7 | 9
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Time to Disease Progression
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to cancer, whichever came first. Tumor progression was determined from oncologic assessment data (where data met the criteria for progressive disease [PD])
Time Frame: Baseline up to end of treatment
Population: A substantial number of participants were not followed-up prior to disease progression, therefore time to disease progression was not estimated.
Arm/Group | CP-751,871 0.025 mg/kg | CP-751,871 0.05 mg/kg | CP-751,871 0.1 mg/kg | CP-751,871 0.2 mg/kg | CP-751,871 0.4 mg/kg | CP-751,871 0.8 mg/kg | CP-751,871 1.5 mg/kg | CP-751,871 3 mg/kg | CP-751,871 6 mg/kg | CP-751,871 10 mg/kg | CP-751,871 20 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- CP-751,871: CP-751,871 0.025, 0.05, 0.1, 0.2, 0.4, 0.8, 1.5, 3 and 6 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks), and dose of 50% from the Cycle 1 dose administered on Day 1 of subsequent cycles, starting from Cycle 2 (4 weeks); CP-751,871 10 and 20 mg/kg administered intravenously on Day 1 of Cycle 1 (4 weeks or 8 weeks) and subsequent cycles, starting from Cycle 2 (4 weeks) (adverse events from all dosing groups were combined as a whole)
Arm/Group | CP-751,871
Serious Adverse Events (participants affected / at risk) | 21/47
Other Adverse Events (participants affected / at risk) | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 (N=47)
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 4
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Chest pain (General disorders) | 1
Muscle hemorrhage (Musculoskeletal and connective tissue disorders) | 1
Disease progression (General disorders) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urosepsis (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Biliary colic (Gastrointestinal disorders) | 1
Cholelithiasis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Fatigue (General disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Asthenia (General disorders) | 4
Hypotension (Cardiac disorders) | 1
Central line infection (Infections and infestations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Speech disorder (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Aggravation reaction (General disorders) | 1
Creatinine increased (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Accidental fall (General disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Myasthenia (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Acute kidney failure (Renal and urinary disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-751,871 (N=47)
ABDOMINAL PAIN (General disorders) | 4
ASTHENIA (General disorders) | 20
CHEST PAIN (General disorders) | 3
HEADACHE (General disorders) | 3
LESION, OTHER AND UNSPECIFIED (General disorders) | 3
PAIN (General disorders) | 6
ANOREXIA (Gastrointestinal disorders) | 4
CONSTIPATION (Gastrointestinal disorders) | 3
DIARRHEA (Gastrointestinal disorders) | 8
DYSPEPSIA (Gastrointestinal disorders) | 7
GINGIVITIS (Gastrointestinal disorders) | 3
NAUSEA (Gastrointestinal disorders) | 9
ANEMIA (Blood and lymphatic system disorders) | 17
HYPOCHROMIC ANEMIA (Blood and lymphatic system disorders) | 4
LEUKOPENIA (Blood and lymphatic system disorders) | 9
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 15
CREATININE INCREASED (Metabolism and nutrition disorders) | 7
DEHYDRATION (Metabolism and nutrition disorders) | 4
HYPERCALCEMIA (Metabolism and nutrition disorders) | 10
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 10
HYPERKALEMIA (Metabolism and nutrition disorders) | 3
HYPERPHOSPHATEMIA (Metabolism and nutrition disorders) | 4
HYPERURICEMIA (Metabolism and nutrition disorders) | 7
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3
HYPONATREMIA (Metabolism and nutrition disorders) | 3
SGOT INCREASED (Metabolism and nutrition disorders) | 9
SGPT INCREASED (Metabolism and nutrition disorders) | 5
WEIGHT LOSS (Metabolism and nutrition disorders) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7
BONE NECROSIS (Musculoskeletal and connective tissue disorders) | 4
BONE PAIN (Musculoskeletal and connective tissue disorders) | 5
LEG CRAMPS (Musculoskeletal and connective tissue disorders) | 5
MYASTHENIA (Musculoskeletal and connective tissue disorders) | 6
ANXIETY (Nervous system disorders) | 3
DIZZINESS (Nervous system disorders) | 4
INSOMNIA (Nervous system disorders) | 5
MUSCULAR HYPERTONIA (Nervous system disorders) | 4
NEUROPATHY (Nervous system disorders) | 3
TREMOR (Nervous system disorders) | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 4
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 3
RESPIRATORY TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 5
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 3
RASH (Skin and subcutaneous tissue disorders) | 3
SWEATING (Skin and subcutaneous tissue disorders) | 3
ABNORMAL VISION (Eye disorders) | 3
URINARY TRACT INFECTION (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.